CLINICAL TRIAL: NCT01012284
Title: Pharmacokinetics, Safety, and Tolerability of TMC207 in Subjects With Moderately Impaired Hepatic Function
Brief Title: A Study of TMC207 in Patients With Moderately Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR007501; TMC207-TiDP13-C112 (Other: Tibotec-Virco Virology BVBA); 2009-016437-99 (EudraCT Number)
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Moderate Hepatic Impairment
Keywords: Moderate Hepatic Impairment; Tuberculosis; TMC207; Mycobacterial adenosine triphosphate (ATP)-synthase
MeSH Terms: conditions — Tuberculosis | interventions — bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panel A (Experimental): 8 patients with moderate hepatic impairment classified as moderate as per the Child Pugh Classification.
  Interventions: Drug: TMC207
- Panel B (Experimental): 8 healthy participants who will match to patients with hepatic impairment in Panel A with regards to sex, age (more or less to 5 years), and body mass index.
  Interventions: Drug: TMC207

INTERVENTIONS:
Drug: TMC207 — 400 mg (4 tablets of 100 mg) of TMC207 will be administered as a single dose on Day 1 of the treatment period to participants of both the Panels (Panel A and Panel B)
  Other Names: R207910

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (what the body does to the medication), safety and tolerability of TMC207 and its N-monodesmethyl metabolite (M2) in healthy participants and in patients with moderate hepatic impairment after administration of a single 400 mg dose of TMC207.

DETAILED DESCRIPTION:
This is a Phase I, open label (all people know the identity of the intervention) study of TMC207. The study consists of a screening period and a 4-weeks treatment period. Sixteen participants will be enrolled in two panels. Panel A will include 8 patients of moderate hepatic impairment and Panel B will include 8 healthy participants. Safety evaluations including adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination will be monitored throughout the study. The entire study duration for each participant will be approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* For healthy participant Panel A: Healthy on the basis of physical examination, medical history, vital signs, electrocardiogram and clinical laboratory tests performed at screening
* Should match to a patient with hepatic impairment with regards to sex, age (more or less to 5 years), and body mass index
* For patients in Panel B with moderate hepatic impairment: history of hepatic disease, documented liver cirrhosis and moderate liver function impairment defined by the Child-Pugh classification

Exclusion Criteria:

* A positive tuberculin skin test indicating latent tuberculosis
* A positive human immunodeficiency virus (HIV)-1 or HIV-2 test at screening
* Moderate hepatic impairment patients with acute hepatitis, Hepatic carcinoma, Grade 3 or 4 encephalopathy, or active candidate for liver transplantation
* Matched healthy participants with current active hepatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of TMC207 | 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, 672 hours
Time to reach the maximum plasma concentration of TMC207 | 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, 672 hours
Area under curve from time of administration up to 72 hours post dosing of TMC207 | 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, 672 hours
Area under curve from time of administration up to the last time point with a measurable concentration post dosing of TMC207 | 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, 672 hours
Area under curve extrapolated to infinity of TMC207 | 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, 672 hours
Maximum plasma concentration of N-monodesmethyl metabolite | 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, 672 hours
Time to reach the maximum plasma concentration of N-monodesmethyl metabolite | 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, 672 hours
Area under curve from time of administration up to 72 hours post dosing of N-monodesmethyl metabolite | 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, 672 hours
Area under curve from time of administration up to the last time point with a measurable concentration post dosing of N-monodesmethyl metabolite | 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, 672 hours
Area under curve extrapolated to infinity of N-monodesmethyl metabolite | 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, 672 hours

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | up to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA

REFERENCES:
- See also: An Open-Label, Prospective, Non-Comparative Study to Evaluate the Efficacy and Safety of Paliperidone Palmitate in Subjects With Acute Schizophrenia. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1632&filename=CR007501_CSR.pdf.pdf